CLINICAL TRIAL: NCT01463124
Title: School Nurse Intervention and After School Exercise Program for Overweight Teens
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Lori Pbert, Professor of Medicine, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21HL110208 (NIH)
Record Dates: First submitted 2011-10-24; First posted 2011-11-01 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Overweight; Obesity
Keywords: School Nurse; Overweight; Obesity; Counseling; Intervention; Exercise
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lookin' Good Feelin' Good (Experimental): Six 30-minute individual student-centered counseling sessions delivered by school nurses during the first two months followed by weekly weigh-ins and monthly visits over the subsequent 6 months, plus an exercise program in the school 3 times a week for the full eight months of the intervention.
  Interventions: Behavioral: Lookin' Good Feelin' Good
- Information attention-control (Active Comparator): Six individual sessions with school nurse over the first two months followed by monthly visits over the remaining 6 months to check weight and behavior changes and provide a series of pamphlets on weight and weight management.
  Interventions: Behavioral: Information attention-control

INTERVENTIONS:
Behavioral: Lookin' Good Feelin' Good — Six 30-minute individual student-centered counseling sessions delivered by school nurses during the first two months followed by weekly weigh-ins and monthly visits over the subsequent 6 months, plus an exercise program in the school 3 times a week for the full eight months of the intervention.
  Arms: Lookin' Good Feelin' Good
Behavioral: Information attention-control — Six individual sessions with school nurse over the first two months followed by monthly visits over the remaining 6 months to check weight and behavior changes and provide a series of pamphlets on weight and weight management.
  Arms: Information attention-control

SUMMARY:
Adolescent overweight and obesity have increased dramatically in the past several decades. High schools are well-positioned to deliver weight loss treatment to overweight and obese adolescents, as they have the facilities and staff to deliver a physical activity program, school nurses with the skills to provide counseling, and are easily accessible by adolescents. This exploratory study will test the feasibility and ability of a school-based intervention, consisting of school nurse counseling and a school-based exercise program, to reduce BMI and improve dietary quality, physical activity, and sedentary behaviors in overweight and obese adolescents. If effective, this could prove to be a cost-effective and relatively easy intervention to disseminate widely for significant public health impact.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in grades 9 - 12
* BMI > 85th percentile for age/sex
* able to understand and participate in the study
* able and willing to provide informed assent (adolescent) and consent (parent)
* English-speaking with at least one English-speaking parent

Exclusion Criteria:

* planning to move out of the area within the next 8 months
* medical condition that precludes adherence to study dietary recommendations (e.g., pregnancy, Crohn's disease, ulcerative colitis)
* diagnosis of a serious psychiatric illness (e.g., psychiatric hospitalization, eating disorder, suicidal) within the past 5 years
* genetic or endocrine causes of obesity (e.g., pradi Willi, Cushing's Syndrome)
* developmental delay that would prevent participation in the intervention or measurements
* prescribed medications associated with weight gain (e.g.,oral steroids)
* morbidly obese, defined as weighing > 300 pounds

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 126 (Actual)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | One academic year (8 months)
  Lookin Good Feelin Good (LGFG) program participants will achieve greater reduction in BMI z-scores than Information attention control (IC) participants after one academic year (8 months) of intervention
Participation in exercise program | One academic year (8 months)
  LGFG participants will report greater than 90% adherence to intervention protocol by school nurses on Patient Exit Interview (PEI) checklists following each of the 6 visits and will attend at least 75% of the exercise sessions.

SECONDARY OUTCOMES:
Self-management | One academic year (8 months)
  LGFG participants will report greater improvements in dietary quality, physical activity and sedentary behavior than IC participants at 8 month follow-up, as measured by 24-hour dietary recall (24HDR), accelerometers, and measures of specific diet, physical activity and sedentary behaviors targeted by the intervention. Improvements will mediate the relationship between condition and BMI.
Physiologic outcomes | One academic year (8 months)
  To evaluate the effect of the LGFG compared to IC condition on changes in secondary physiologic outcomes, including waist circumference, estimate of body fat, and blood pressure.
Psychosocial outcomes | One academic year (8 months)
  To evaluate the effect of the LGFG compared to the IC condition on changes in psychosocial outcomes including self-efficacy, quality of life, and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Pbert, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States